CLINICAL TRIAL: NCT01236950
Title: Study of an Essential Oil and a Delmopinol Mouthrinse Effect on Dental Plaque Accumulation Index, Gingivitis Index and on Streptococcus Mutans, Lactobacillus, Aerobic and Anaerobic Oral Bacteria Colony Counts.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: Instituto Piaget (Other)
Responsible Party: Henrique Soares Luis, Faculdade de Medicina Dentária da Universidade de Lisboa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9/2006a
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-07

CONDITIONS: Gingivitis; Dental Plaque Accumulation
Keywords: Clinical Trial; Prevention Mouthrinse
MeSH Terms: conditions — Gingivitis | interventions — delmopinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Delmopinol mouthrinse (Experimental): Subjects use the delmopinol mouthrinse
  Interventions: Drug: Delmopinol mouthrinse
- Control (No Intervention): Subjects with no use of mouthrinse
- Essential oils mouthrinse (Experimental): Subjects using the essential oils mouthrinse
  Interventions: Drug: Essential oils mouthrinse

INTERVENTIONS:
Drug: Essential oils mouthrinse — Commercial mouthrinse with manufacturer's use indication
  Other Names: Listerine Cool Mint
  Arms: Essential oils mouthrinse
Drug: Delmopinol mouthrinse — Commercial mouthrinse with manufacturer's use indication
  Other Names: Decapinol
  Arms: Delmopinol mouthrinse

SUMMARY:
The use of mouthrinses may be of relevance as a complement to daily dental hygiene procedures, especially for patients who do not comply with a proper mechanical removal of dental plaque. Essential oils and delmopinol mouthrinses are effective to reduce dental plaque accumulation and gingivitis. Also an effect on dental bacteria can be found. The study hypothesis states that there are no differences between the mouthrinses on the reduction of gingivitis and dental plaque accumulation as well on the bacterial counts of Streptococcus mutans, Lactobacillus, aerobic and anaerobic bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the dental hygiene clinic of Faculdade de Medicina Dentária
* Signature of consent form
* Have, at least, two quadrant with 6 teeth each
* Gingival Index at baseline less than 3
* Presence of dental plaque

Exclusion Criteria:

* Use of a mouthrinse
* Dental Hygiene appointment in the past 6 months
* Use of antibiotics in teh past 3 months
* Presence of extensive caries and fractures of teeth

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Loe & Silness Gingival Index (1963) | change from baseline in gingival index at two weeks
  data collected at the begining of the study and two weeks after mouthrinse usage.
Quigley, Hein & Turesky Dental Plaque Index (1970) | change from baseline in plaque index at two weeks
  data collected at the begining of the study and two weeks after mouthrinse usage.

SECONDARY OUTCOMES:
Streptococcus mutans CFU | change from baseline in CFU counts at two weeks
  data collected at the begining of the study and two weeks after mouthrinse usage.
Lactobacillus CFU | change from baseline in CFU counts at two weeks
  data collected at the begining of the study and two weeks after mouthrinse usage.
Aerobic and anaerobic oral bacteria CFU | change from baseline in CFU counts at two weeks
  data collected at the begining of the study and two weeks after mouthrinse usage.

CONTACTS AND LOCATIONS:
Overall Officials: Mario F Bernardo, PhD, Study Director — Faculdade de Medicina Dentária da Universidade de Lisboa
Locations (1):
- Faculdade de Medicina Dentária da Universidade de Lisboa, Lisbon, Lisbon District, Portugal

REFERENCES:
- [Background] Abbott DM, Gunsolley JC, Koertge TE, Payne EL. The relative efficacy of 0.1% and 0.2% delmopinol mouthrinses in inhibiting the development of supragingival dental plaque and gingivitis in man. J Periodontol. 1994 May;65(5):437-41. doi: 10.1902/jop.1994.65.5.437. PMID 8046559
- [Background] Addy M, Moran J, Newcombe RG. Meta-analyses of studies of 0.2% delmopinol mouth rinse as an adjunct to gingival health and plaque control measures. J Clin Periodontol. 2007 Jan;34(1):58-65. doi: 10.1111/j.1600-051X.2006.01013.x. Epub 2006 Nov 20. PMID 17116159
- [Background] Baehni PC, Takeuchi Y. Anti-plaque agents in the prevention of biofilm-associated oral diseases. Oral Dis. 2003;9 Suppl 1:23-9. doi: 10.1034/j.1601-0825.9.s1.5.x. PMID 12974527
- [Background] Barnett ML. The rationale for the daily use of an antimicrobial mouthrinse. J Am Dent Assoc. 2006 Nov;137 Suppl:16S-21S. doi: 10.14219/jada.archive.2006.0408. PMID 17035671
- [Background] Fine DH, Furgang D, Barnett ML, Drew C, Steinberg L, Charles CH, Vincent JW. Effect of an essential oil-containing antiseptic mouthrinse on plaque and salivary Streptococcus mutans levels. J Clin Periodontol. 2000 Mar;27(3):157-61. doi: 10.1034/j.1600-051x.2000.027003157.x. PMID 10743861
- [Background] Gordon JM, Lamster IB, Seiger MC. Efficacy of Listerine antiseptic in inhibiting the development of plaque and gingivitis. J Clin Periodontol. 1985 Sep;12(8):697-704. doi: 10.1111/j.1600-051x.1985.tb00941.x. PMID 3902908
- [Background] Ouhayoun JP. Penetrating the plaque biofilm: impact of essential oil mouthwash. J Clin Periodontol. 2003;30 Suppl 5:10-2. doi: 10.1034/j.1600-051x.30.s5.4.x. PMID 12787196